CLINICAL TRIAL: NCT04190186
Title: Hybrid Ablation Plus Medical Therapy for Persistent Atrial Fibrillation (HYBRID AF)
Brief Title: Hybrid Ablation Plus Medical Therapy for Persistent Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Biotronik, Inc. (Industry)
Responsible Party: Principal Investigator, David Huang, Professor Medicine M&D-Cardiology Div, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00004318
Record Dates: First submitted 2019-11-20; First posted 2019-12-09 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Biotronik BioMonitor; ICM; AF Ablation; Atrial arrhythmia
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Biotronik ICM-guided AF management (Active Comparator): ICM obtained data will be actively used to guide and monitor treatment .
  Interventions: Device: Insertable Cardiac Monitor
- Conventional AF Management (No Intervention): Treating physicians/nurses will be blinded to the AF episodes data from the monitor, but will be provided information on asystole, or ventricular arrhythmia events (for safety).

INTERVENTIONS:
Device: Insertable Cardiac Monitor — Implantable device that provides accurate daily transmission of cardiac electrical data for arrhythmia detection.
  Other Names: BioMonitor3® or future generation of Biotronik ICM
  Arms: Biotronik ICM-guided AF management

SUMMARY:
This clinical trial is designed to compare two management strategies for the treatment of asymptomatic/subclinical atrial fibrillation after ablation based on data from the Biotronik ICM (BioMonitor3® or future generation of Biotronik ICM).

DETAILED DESCRIPTION:
In this study, subjects will be randomized (1:1) to conventional AF management vs. Biotronik ICM-guided AF management following ablation for persistent AF. Subjects will be followed for 15 months including a 3 month blanking period following AF ablation. The study subject population will include subjects with persistent atrial fibrillation (sustained AF episode lasting more than 7 days, but less than 1 year), according to current guideline indications for persistent AF ablation and ICM (Biotronik ICM) implantation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* History of persistent atrial fibrillation (sustained AF episode lasting more than 7 days, but less than a year)
* Planned to undergo first AF ablation with successful Biotronik ICM implant before or at time of ablation

Exclusion Criteria:

* Paroxysmal atrial fibrillation
* Long persistent atrial fibrillation (continuous atrial fibrillation that lasts more than 1 year)
* Permanent atrial fibrillation
* Left atrial diameter of 60 mm or greater
* Patients with CHF status prohibiting EP study and ablation, but may be re-considered for enrollment later after effective treatment
* Patients with metabolic derangements (e.g. renal/hepatic failure, electrolyte disturbance, etc.), prohibiting EP study and ablation or antiarrhythmic medical therapy (e.g. dofetilide, sotalol or amiodarone, etc.)
* Patients with an intra-cardiac thrombus, but may be re-considered for enrollment later after effective treatment
* Serious known concomitant disease with a life expectancy of < 1 year
* Pregnancy or nursing
* Unwilling or unable to give informed consent
* Existing CIED such as pacemaker or ICD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Huang, MD, Principal Investigator — University of Rochester
Locations (4):
- United States (4):
  - Michigan Heart, PC, Ypsilanti, Michigan
  - Cardiology Associates Research, LLC, Tupelo, Mississippi
  - Rochester Regional Health, Rochester, New York
  - University of Rochester, Rochester, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verma A, Jiang CY, Betts TR, Chen J, Deisenhofer I, Mantovan R, Macle L, Morillo CA, Haverkamp W, Weerasooriya R, Albenque JP, Nardi S, Menardi E, Novak P, Sanders P; STAR AF II Investigators. Approaches to catheter ablation for persistent atrial fibrillation. N Engl J Med. 2015 May 7;372(19):1812-22. doi: 10.1056/NEJMoa1408288. PMID 25946280
- [Background] Huang DT, Monahan KM, Zimetbaum P, Papageorgiou P, Epstein LM, Josephson ME. Hybrid pharmacologic and ablative therapy: a novel and effective approach for the management of atrial fibrillation. J Cardiovasc Electrophysiol. 1998 May;9(5):462-9. doi: 10.1111/j.1540-8167.1998.tb01837.x. PMID 9607453
- [Background] Kirchhof P, Calkins H. Catheter ablation in patients with persistent atrial fibrillation. Eur Heart J. 2017 Jan 1;38(1):20-26. doi: 10.1093/eurheartj/ehw260. Epub 2016 Jul 7. PMID 27389907
- [Background] Willems S, Khairy P, Andrade JG, Hoffmann BA, Levesque S, Verma A, Weerasooriya R, Novak P, Arentz T, Deisenhofer I, Rostock T, Steven D, Rivard L, Guerra PG, Dyrda K, Mondesert B, Dubuc M, Thibault B, Talajic M, Roy D, Nattel S, Macle L; ADVICE Trial Investigators*. Redefining the Blanking Period After Catheter Ablation for Paroxysmal Atrial Fibrillation: Insights From the ADVICE (Adenosine Following Pulmonary Vein Isolation to Target Dormant Conduction Elimination) Trial. Circ Arrhythm Electrophysiol. 2016 Aug;9(8):e003909. doi: 10.1161/CIRCEP.115.003909. PMID 27516462
- [Background] Schreiber D, Rostock T, Frohlich M, Sultan A, Servatius H, Hoffmann BA, Luker J, Berner I, Schaffer B, Wegscheider K, Lezius S, Willems S, Steven D. Five-year follow-up after catheter ablation of persistent atrial fibrillation using the stepwise approach and prognostic factors for success. Circ Arrhythm Electrophysiol. 2015 Apr;8(2):308-17. doi: 10.1161/CIRCEP.114.001672. Epub 2015 Mar 5. PMID 25744570
- [Background] Reiffel JA, Camm AJ, Belardinelli L, Zeng D, Karwatowska-Prokopczuk E, Olmsted A, Zareba W, Rosero S, Kowey P; HARMONY Investigators. The HARMONY Trial: Combined Ranolazine and Dronedarone in the Management of Paroxysmal Atrial Fibrillation: Mechanistic and Therapeutic Synergism. Circ Arrhythm Electrophysiol. 2015 Oct;8(5):1048-56. doi: 10.1161/CIRCEP.115.002856. Epub 2015 Jul 30. PMID 26226999
- [Background] Tondo C, Iacopino S, Pieragnoli P, Molon G, Verlato R, Curnis A, Landolina M, Allocca G, Arena G, Fassini G, Sciarra L, Luzi M, Manfrin M, Padeletti L; ClinicalService 1STOP Project Investigators. Pulmonary vein isolation cryoablation for patients with persistent and long-standing persistent atrial fibrillation: Clinical outcomes from the real-world multicenter observational project. Heart Rhythm. 2018 Mar;15(3):363-368. doi: 10.1016/j.hrthm.2017.10.038. Epub 2017 Oct 26. PMID 29107190

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Biotronik ICM-guided AF Management | Conventional AF Management
Started | 27 | 28
Completed | 20 | 20
Not Completed | 7 | 8
Not completed — ILR is no longer functioning | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Subject choice to explant | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Study was stopped | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biotronik ICM-guided AF Management | Conventional AF Management | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 21 | 37
  >=65 years | 11 | 7 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.7 (8.4) | 63.5 (9.3) | 64.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 17 | 22 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 27 | 28 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: Atrial Fibrillation (AF) Burden Defined as the Mean Amount of Time Spent in AF Over a Pre-specified Period of Time (Excluding Short AF Episodes of ≤30 Seconds) by the Biotronik ICM (BioMonitor3® or Future Generation of Biotronik ICM).
Description: In the present study AF burden will be assessed at 3-month intervals during the 12 months following the blanking period (3-months post-ablation), and the difference at the end of the follow-up period of one year will serve as the primary comparison outcome between the two treatment groups.
Time Frame: Between months 3 and 15 after the ablation procedure (to exclude the first 3 month blanking period)
Measure: Mean (Standard Deviation); unit: percentage of time spent in AF
Arm/Group | Biotronik ICM-guided AF Management | Conventional AF Management
Number analyzed (Participants) | 27 | 28
percentage of time spent in AF | 4.99 (8.26) | 2.57 (4.41)
Statistical Analysis 1: Comparison: Biotronik ICM-guided AF Management vs Conventional AF Management; Test type: Superiority; p = 0.594, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.49

2. Secondary Outcome: Number of Participants With Clinically Significant (>30 Min) Atrial Arrhythmia (Atrial Fibrillation, Atrial Flutter or Atrial Tachycardia) as Detected and Documented by Biotronik ICM After the Performance of the Index AF Ablation Procedure.
Time Frame: Between enrollment and 15 months (excluding the initial 3-month blanking period) (assessed in a recurrent event analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | Biotronik ICM-guided AF Management | Conventional AF Management
Number analyzed (Participants) | 27 | 28
Participants | 0.0 | 0.0

3. Secondary Outcome: Number of Participants With Symptomatic AF Recurrence (Regardless of Duration).
Time Frame: Between enrollment and 15 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Biotronik ICM-guided AF Management | Conventional AF Management
Number analyzed (Participants) | 27 | 28
Participants | 0.0 | 0.0

4. Secondary Outcome: Number of Participants With Repeat AF Ablation.
Time Frame: Between enrollment and 15 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Biotronik ICM-guided AF Management | Conventional AF Management
Number analyzed (Participants) | 27 | 28
Participants | 3.0 | 4.0

5. Secondary Outcome: Number of Participants With Cardiac Hospitalization.
Time Frame: Between enrollment and 15 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Biotronik ICM-guided AF Management | Conventional AF Management
Number analyzed (Participants) | 27 | 28
Participants | 3 | 3

6. Secondary Outcome: Number of Deaths.
Time Frame: Between enrollment and 15 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Biotronik ICM-guided AF Management | Conventional AF Management
Number analyzed (Participants) | 27 | 28
Participants | 0 | 0

7. Secondary Outcome: Number of Participants With Healthcare Utilization, Defined as Hospitalization for Any Cause, ED Visits, and Unplanned Office Visits.
Time Frame: Between enrollment and 15 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Biotronik ICM-guided AF Management | Conventional AF Management
Number analyzed (Participants) | 27 | 28
Participants | 5 | 7

8. Secondary Outcome: Number of Participants With Atrial Flutter or Tachycardia.
Description: Incidence of atrial flutter or tachycardia after the index ablation procedure
Time Frame: Between months 3 and 15 after the ablation procedure (to exclude the first 3 month blanking period)
Measure: Count of Participants; unit: Participants
Arm/Group | Biotronik ICM-guided AF Management | Conventional AF Management
Number analyzed (Participants) | 27 | 28
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With Incidence of Repeat Procedures.
Time Frame: Between months 3 and 15 after the ablation procedure (to exclude the first 3 month blanking period)
Measure: Count of Participants; unit: Participants
Arm/Group | Biotronik ICM-guided AF Management | Conventional AF Management
Number analyzed (Participants) | 27 | 28
Participants | 5 | 4

10. Secondary Outcome: Number of Participants With Major Adverse Events Requiring Rehospitalization During Follow-up.
Time Frame: Between months 3 and 15 after the ablation procedure (to exclude the first 3 month blanking period)
Measure: Count of Participants; unit: Participants
Arm/Group | Biotronik ICM-guided AF Management | Conventional AF Management
Number analyzed (Participants) | 27 | 28
Participants | 2 | 3

11. Secondary Outcome: Quality of Life as Assessed by the Atrial Fibrillation Effect on QualiTy-of-life (AFEQT) Questionnaire
Description: The Atrial Fibrillation Effect on Quality-of-Life (AFEQT) questionnaire is a validated, disease-specific instrument used to assess quality of life in individuals with atrial fibrillation. It includes 20 questions across four domains: Symptoms, Daily Activities, Treatment Concern, and Treatment Satisfaction.
  The AFEQT provides both domain-specific scores and an overall total score. Scores for each domain and the Total Score range from 0 to 100. Higher scores indicate better quality of life, with 100 representing no symptoms or limitations and 0 representing severe symptoms or limitations. The Total Score is calculated by averaging the scores from the three core domains (Symptoms, daily activities, and treatment concern).
Time Frame: Between months 3 and 15 after the ablation procedure (to exclude the first 3 month blanking period)
Measure: Mean (Standard Deviation); unit: Score (from the AFEQT questionnaire)
Arm/Group | Biotronik ICM-guided AF Management | Conventional AF Management
Number analyzed (Participants) | 27 | 28
Score (from the AFEQT questionnaire) | 88.0 (14.6) | 85.9 (12.6)

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Biotronik ICM-guided AF Management | Conventional AF Management
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 3/27 | 3/28
Other Adverse Events (participants affected / at risk) | 8/27 | 9/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Biotronik ICM-guided AF Management (N=27) | Conventional AF Management (N=28)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Atrial Arrhythmia (Cardiac disorders) | 0 | 1
Congestive Heart Failure (Cardiac disorders) | 1 | 0
Generalized Weakness (General disorders) | 0 | 2
Pain (General) (General disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Biotronik ICM-guided AF Management (N=27) | Conventional AF Management (N=28)
Atrial Fibrillation (Cardiac disorders) | 2 | 1
Cough Increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fever (General disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Atrial Arrhythmia (Cardiac disorders) | 0 | 2
Congestive Heart Failure (Cardiac disorders) | 1 | 0
Generalized Weakness (General disorders) | 0 | 2
Pain (General) (General disorders) | 3 | 1
Pericarditis (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT04190186/Prot_SAP_000.pdf